CLINICAL TRIAL: NCT05103345
Title: A Phase I/IIa, Open-label, Dose Escalation and Dose-Expansion Study to Evaluate the Safety and Tolerability of Modified Salmonella Typhimurium SGN1 Administered Via Intratumoral Injection in Patients With Advanced Solid Tumors
Brief Title: Study of SGN1 Administered Via Intratumoral Injection in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Sinogen Pharmaceutical Co., Ltd (Other)
Collaborators: Pharmaron (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN-P01-002
Record Dates: First submitted 2021-09-24; First posted 2021-11-02 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: This study will be conducted in 2 parts: Part 1 is a phase I open-label, dose escalation study phase. Part 2 is as a part of a phase Ib/IIa study, which is a specific Tumor-type expansion study.
  The standard 3+3 dose escalation algorithm will be applied to explore dose limiting toxicity (DLTs) in at least 4 sequential cohorts with 3- 6 patients and identify the maximally tolerated dose (MTD).
  When the cohort is completed in Part 1, the Part 2 study could be started according to the SMC evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): SGN1 will be injected into the target lesion intratumorally. According to the dose levels, the administered dose will be 0.5×108 CFU, 1×108 CFU, 2×108 CFU, 4×108 CFU, 6×108 CFU (optional). The patient will be administered once every week for 3 consecutive weeks followed by 1-week rest in 28-day treatment cycles. The duration of administration is until isease complete response/inability to continue intratumoral administration or disease progression, or intolerable toxicity or death or voluntary withdrawal or end of study, whichever came first.
  The standard 3+3 dose escalation algorithm will be applied to explore dose limiting toxicity (DLTs) in at least 4 sequential cohorts with 3- 6 patients and identify the maximally tolerated dose (MTD).
  When the cohort is completed in Part 1, the Part 2 study could be started according to the SMC evaluation. Enrollment of 2-4 dose level expansions will be opened to determine the safety and efficacy of SGN1 in specific tumor types
  Interventions: Drug: SGN1

INTERVENTIONS:
Drug: SGN1 — SGN1,will be administered intratumorally,which dosage is 0.9-2.0×109 cfu /vial.
  Other Names: SalMet-Vec

SUMMARY:
Objectives: To characterize safety, tolerability, MTD and OBD of intratumoral injection of SGN1 in patients with advanced solid tumors, and to preliminarily investigate the efficacy and safety of SGN1 in specific tumor subtypes.

Study Rationale: The mechanism of action for SGN1 is based on the fact that most tumors are methionine dependent. SGN1 is designed to be used as a tumor therapeutic bacterium that can preferentially replicate and accumulate in tumors and starve them of essential amino acids by delivering the oncolytic enzyme L-Methioninase.

Patient Population: Patients presenting with histologically confirmed advanced and/or metastatic solid tumors that are refractory to standard therapy and for which no other conventional therapy exists.

DETAILED DESCRIPTION:
Methionine starvation can powerfully modulate DNA methylation, cell cycle transition, polyamines and antioxidant synthesis of tumor cells, in contrast to normal ones. L-Methioninase is a pyridoxal phosphate dependent enzyme that catalyzes the γ-elimination reaction of L-methionine to methanethiol, α-ketobutyrate and ammonia . Absolute-dependency on exogenous supply of L-methionine, not homocysteine, for growth and proliferation of tumors is the pivotal biochemical criterion for various human cancers.

SGN1 is a genetically modified strain of Salmonella enterica, serotype typhimurium that expresses L-Methioninase. The attenuated live bacterium has been investigated in China for utility in treating advanced solid tumors. The mechanism of action for SGN1 is based on the fact that most tumors are methionine dependent. SGN1 is designed to be used as a tumor therapeutic bacterium that can preferentially replicate and accumulate in tumors and starve them of essential amino acids by delivering the oncolytic enzyme L-Methioninase.

This study is a multi-center phase I/IIa clinical trial with 2 parts:

Part 1 is a phase I open-label, dose escalation study phase. The purpose of Part 1 is to characterize safety, tolerability, MTD and OBD of intratumoral injection of SGN1 in patients with advanced solid tumors. Part 2 is as a part of a phase Ib/IIa study, which is a specific Tumor-type expansion study, the purpose of Part 2 is to preliminarily investigate the efficacy and safety of SGN1 in specific tumor subtypes at Safety Monitoring Committee (SMC) determined doses.

SGN1 will be administrated in 28-days cycles (once weekly for 3 weeks followed by 1-week rest). Intratumoral injection of SGN1 can be performed directly using methods including but not limited to color doppler ultrasound guidance, which is the preferred method. If the Investigator(s) judge(s) it necessary, the intratumoral injection can also be performed under CT guidance by an interventional radiologist or specialist with adequate qualifications and trainings.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, patients who have laboratory values outside of the specified ranges will be permitted to be retested. Patients who meet the following criteria at the screening visit will be eligible for participation in the study:

1. Male or female aged 18~75 years((including 18 and 75 years)) at the time of informed consent;
2. Part 1: Patients with advanced stage (unresectable or metastatic) solid tumors including but not limited to small cell lung cancer, non-small cell lung cancer (adeno- and squamous), Hodgkin's lymphoma or non-Hodgkin's lymphoma, sarcoma, cervical carcinoma, Melanoma, head and neck cancer, breast cancer, ovarian cancer, pseudomyxoma peritoneum (Pseudomyxoma peritonei, PMP) and hepatocellular carcinoma characterized by failure of standard treatment (disease progression or intolerance, such as chemotherapy, targeted therapy, and other immunotherapies) or patients who have no standard treatment or patients who are intolerable to standard treatment; Note: For all tumor species included, standard treatment will refer to current Chinese Society of Clinical Oncology (CSCO)/National Comprehensive Cancer Network (NCCN) guidelines.

   Standard treatment failure refers to patients who have disease progression after the existing standard of care recommended by CSCO/NCCN guidelines, or relapse/metastasis after standard of care.

   Non-standard treatment refers to patients who have received the treatment recommended by the guidelines and currently have no other effective treatment options.
3. Part 2: the specific tumor-type expansion study may enroll the following patients: Patients with advanced HNSCC, Sarcoma, HCC, cervical cancer, melanoma, or other tumor type with potential efficacy signal observed in Part 1, who have failed to standard therapy or who are intolerant to the standard treatment.
4. Patients must have the main lesion suitable for local injection of SGN1. The tumors must be in situ or metastatic solid tumors that are subcutaneous, palpable, or can be injected directly using methods including but not limited to color doppler ultrasound guidance, which is the preferred method. If the Investigator(s) judge(s) it necessary, the intratumoral injection can also be performed under CT guidance by an interventional radiologist or specialist with adequate qualifications and trainings, provided that these tumors do not invade the walls of blood vessels or hollow organs confirmed by previous imaging studies and Investigator assessment (no risk of major bleeding or hollow organ perforation).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Life expectancy ≥ 12 weeks.
7. Patients have recovered from any toxic reaction to previous medications (≤Grade 1 based on NCI-CTCAE v 5.0, except

   1. Hair loss;
   2. Pigmentation;
   3. The long-term toxicity caused by radiotherapy and cannot be recovered by the Investigator's judgment;
   4. Platinum induced neurotoxicity of grade 2 and below;
   5. Hemoglobin at 90 ~ 100 g/L (including boundary value) or stable status assessed by the Investigator.
   6. Patients with adrenal and thyroid dysfunction who maintain a stable state after drug treatment as judged by the Investigator may be included in this study; Patients with toxic reactions of single indicator grade 2 or above that with no clinical significance or clinical treatment measures, which will be determined by the investigator if not affect the study, can also be included.
8. At least one measurable injected lesion as determined by RECIST 1.1(for solid tumors).
9. Laboratory tests must meet the following requirements and have not received any blood cell growth factor 14 days before the test and no blood transfusions within 14 days prior to screening (patients with laboratory values outside of the specified ranges will be permitted to be retested during the screening period in order to meet the criteria),

   1. Absolute count of neutrophils (ANC) ≥1.5×109/L, platelet ≥75×109/L; Hemoglobin ≥90 g/L;
   2. Serum albumin ≥ 30 g/L; Bilirubin ≤1.5 × ULN, ALT and AST ≤2.5 × ULN;
   3. In patients with liver metastasis, ALT and AST≤5 × ULN;
   4. Creatinine clearance ≥50 mL/min (standard Cockcroft -Gault formula) or Cr ≤1.5 ×ULN: urinary protein ≤2+ or urinary protein quantitative <1.0 g/L;
   5. International standardized ratio of coagulation function (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (if the patient is taking concomitant anticoagulant medication, whether the coagulation function is qualified will be determined by the Investigator).
10. If female, be either postmenopausal for at least 1 year with documented follicle stimulating hormone (FSH) >30 IU/L, or surgically sterile for at least 3 months, or if a woman of childbearing potential, must be non-pregnant confirmed by blood and urine pregnancy tests, and non-lactating.
11. Female patients of childbearing potential must agree to use acceptable method(s) of contraception from consent through at least 6 months after the last dose of drug intratumoral injection.
12. Male patients of reproductive capacity must agree to use effective contraception from start of mobilization through at least 6 months after the last dose of drug intratumoral injection.
13. Patients must be able to follow up after the treatment.
14. Patients must understand and voluntarily sign the informed consent form.

Exclusion Criteria

Patients will be excluded from participation of the study for any of the following criteria:

1. Prior treatment with oncolytic bacteria viral or anti-tumor bacteria therapy.
2. Patients with extremely large tumor (the longest diameter of a single tumor does not exceed 8 cm in principle); patients with multiple lesions cannot receive intratumoral injection, it mainly refers to patients with extensive metastasis who are not suitable for local treatment;
3. Patients who are allergic or intolerant to salmonella sensitive antibiotics, and have infectious diseases and are currently using antibiotics.
4. Present assessable tumors in hollow organs (stomach, esophagus, intestine, urinary tract etc.).
5. Patients who are known to be allergic to the investigational drug or any of its excipients; or rescue medications; or have a severe allergic reaction to other monoclonal antibodies.
6. Patients who have received the following treatments or drugs before the first treatment with the investigational drug:

   1. Major surgery performed within 28 days before the first treatment with the investigational drug (biopsy is allowed for diagnostic purposes);
   2. Immunosuppressive drugs have been administered within 14 days before the first treatment with the investigational drug (Prednisone >10 mg/day, or equivalent doses of corticosteroids), excluding corticosteroid nasal sprays and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e., prednisone not exceeding 10 mg/d or equivalent physiological doses of other corticosteroids);
   3. Inoculation of (attenuated) live virus vaccine: within 28 days before the first dosing of study drug, or during the study period or 60 days after the last dose of study drug; Except for administration of inactivated vaccines and RNA vaccines (e.g., inactivated influenza vaccines and COVID-19 RNA vaccines);
   4. Any anti-tumor therapies (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy or tumor embolization) within 28 days before the first dosing of the investigational drug (if nitrosourea or mitomycin chemotherapy the interval between end of chemotherapy and first dose of study treatment must be no less than 6 weeks).
7. Patients with known uncontrollable or symptomatic active CNS metastases, manifested by clinical symptoms, brain edema, spinal cord compression, cancerous meningitis, leptomeningeal disease, and/or progressive growth. Patients with a history of metastases to the central nervous system or spinal cord compression can be included in the study if they have clearly received treatment and have shown stable clinical manifestations after the discontinuation of anticonvulsants and steroids for 4 weeks before the first dose of the investigational drug.
8. Present with diverticulitis that may cause anaerobic bacteria to multiply or conditions at screening that might promote the unintentional growth of anaerobic bacteria in nontarget lesions.
9. Symptomatic, advanced patients whose tumors have spread to the internal organs and are at risk of life-threatening complications in the short term (including patients with uncontrollable large amounts of effusion (thoracic cavity, pericardial cavity, or abdominal cavity);
10. Patients with any active autoimmune diseases or a history of any autoimmune disease with predictable recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [only patients whose condition can be controlled by hormone replacement therapy can be included]; Patients with skin diseases that do not require systemic treatment such as vitiligo, psoriasis, hair loss, Type I diabetes mellitus, or those with childhood asthma which has been completely relieved and requires no interventions in adulthood, can be included. Those with asthma who need bronchodilators for medical intervention cannot be included);
11. Patients with other active malignant tumor(s) within 2 years before entering the study. Patients with history of cervical carcinoma in situ, superficial or non-invasive bladder cancer or basal cell or squamous cell cancer in situ previously treated with curative intent may be included at the judgment of the Investigator.
12. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as: hepatitis B virus surface antigen [HbsAg] testing positive, HBV-DNA ≥ 500 IU/mL and abnormal liver function; hepatitis C, defined as: hepatitis C antibody [HCV-Ab] testing positive, higher HCV-RNA than the lower limit of detection of the analysis method and abnormal liver function) or hepatitis B and hepatitis C co-infection;
13. Existing cardiac clinical symptoms or diseases that cannot be well controlled, such as:

    1. NYHA grade 2 or above heart failure;
    2. Unstable angina pectoris;
    3. Myocardial infarction occurred within 1 year;
    4. Patients with supraventricular or ventricular arrhythmias that have clinical significance and need treatment or intervention;
    5. Uncontrolled hypertension (systolic blood pressure) ≥160 mmHg and (diastolic blood pressure) ≥100 mmHg after drug treatment;
    6. Patients with valvular heart disease or mitral valve prolapse, aortic valve disease or other source of turbulent cardiac blood flow.
14. Patients with active or uncontrolled infection or fever > 38.5°C of unknown cause or before the first administration of the study drug;
15. Documented salmonella infection within 6 months.
16. Known history of allogeneic organ transplant or allogeneic hematopoietic stem cell transplant.
17. Patients participating in other clinical studies or participating in other clinical studies within 4 weeks or 5 half-lives of other study drugs, whichever is longer, prior to enrollment and receiving experimental drug administration.
18. Known history of psychotropic drug abuse or recreational drug abuse;
19. In the judgment of the Investigator, there are other factors that may lead to termination: for example, adrenal cortex insufficiency, pituitary insufficiency after treatment, and other serious diseases (including mental diseases) need to be treated together, there are serious abnormalities in laboratory examination, family or social factors, which may affect the safety of the patients or test data and sample collection.
20. Patients with implants such as pacemakers, prosthetic cardiac valves, or vascular stents who require long-term anticoagulant therapy;
21. In the Investigator's judgment, patients who are not suitable for other reasons;
22. Abdominal standing position plain film or abdominal CT indicates the possibility of bowel obstruction within 6 months from screening, or the Investigator believes there is a risk of bowel obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From receiving study drug and throughout the study, until 28 days after the last dosing
  An AE is any untoward medical occurrence in a patient or clinical investigation patient, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Events meeting the definition of an AE include:
  * Any abnormal laboratory test results (hematology, serum chemistry, or urinalysis) or other safety assessments (e.g., ECGs, vital signs measurements), including those that worsen from baseline, and was felt to be clinically significant in the medical and scientific judgment of the Investigator.
  * Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
  * New conditions detected or diagnosed after study treatment administration even though it may have been present prior to the start of the study.
  * Signs, symptoms, or the clinical sequelae of a suspected interaction.
Incidence of SAEs | From receiving study drug and throughout the study, until 28 days after the last dosing
  An AE or suspected adverse reaction is considered "serious" if it results in any of the following outcomes:
  * Death
  * Life-threatening
  * In patient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  * Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.
Objective response rate (ORR) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS.
  • The ORR is defined as the proportion of patients who achieve PR or better according to the RECIST v1.1. mRECIST is used to assess Hepatocellular carcinoma only, Choi criteria is used for all solid tumors, during the whole study, as the only exploratory tumor assessment method in the study, and LYRIC is used to assess Lymphoma as assessed by the investigator.
Disease control rate (DCR) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS.
  • The DCR is defined as the proportion of patients who achieve SD or better according to the RECIST v1.1, mRECIST is used to assess Hepatocellular carcinoma only, Choi criteria is used for all solid tumors, during the whole study, as the only exploratory tumor assessment method in the study, and LYRIC is used to assess Lymphoma as assessed by the investigator.
Progression Free Survival (PFS) | From signing the informed consent form until 28 days after the last dose.
  The efficacy endpoints include ORR, DCR and PFS.
  • PFS is defined as the time interval from date of first dose of SGN1 to the date of documented disease progression (iRECIST is used when the patient is suspected to be pseudo disease progression) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days post first dose
  Any of the following judged to be associated with SGN1 may be considered a DLT:
  1. Any Grade 5 adverse event that is at least possibly related to investigational drug
  2. Non-hematological toxicities:
     1. Grade 4 non-hematological toxicities (excluding alopecia) lasting > 3 days despite optimal supportive care (OSC).
     2. Grade 3 non-hematologic toxicities lasting > 7 days despite OSC.
  3. Hematological toxicities:
     1. Grade 4 hematologic toxicities lasting > 7 days (except following b and c).
     2. Grade 3 or 4 febrile neutropenia (body temperature ≥38.5°C) lasting > 7 days.
     3. Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia.
SGN1 level in blood for PK analysis | Before and after SGN1 injection in the first two cycles in Part 1 and Part 2.
  In Part 1 and Part 2, blood sampling will be collected for pharmacokinetics (PK).
  The blood collection times for PK are within 30 minutes predose and 30 minutes postdose of intratumoral injection on C1D1(cycle1 day1), C1D8(cycle1 day8), C1D15(cycle1 day15), C2D1(cycle2 day1), C2D8(cycle2 day8), and C2D15(cycle2 day15), and at the following timepoints after the end of dose on C1D1 and C2D1: 5 minutes (± 1 minute), 10 minutes (± 1 minute), 1 hour (± 2 minutes), 1.5 hours (± 2 minutes), 2 hours (± 2 minutes), 4 hours (± 5 minutes), 6 hours (± 10 minutes), 8 hours (± 15 minutes), 24 hours ± 1 hour, 48 hours ± 1 hour, 72 hours ± 1 hour. If there are still symptoms of fever or infection after 72 hours, extend the PK collection time and expect to increase it every 24 hours(± 1 hour) until the infection symptoms disappear.
Immunogenicity (anti-drug antibodies) | Before and after SGN1 injection in the first 4 cycles in Part 1 and Part 2.
  Anti-drug antibody blood sample collection time points: each predose (within 2 days) in the first 2 cycles, before the first dose in Cycles 3 and 4 (within 2 days), and at the EOT/withdrawal visit.
SGN1 level in blood for bacterial shedding. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 2,blood samples will be collected for Bacterial Shedding.
  Blood samples will be collected within 2 hours prior to the start of SGN1 intratumoral injection on C1D8 and C1D15, and within 24±3 hours after the end of each SGN1 intratumoral injection on C1D8 and C1D15.
  Blood bacterial samples within 30 minutes predose and 30 minutes postdose of intratumoral injection on C1D1, C1D8, C1D15, C2D1, C2D8, and C2D15 are measured in the PK analysis described above. The results from PK blood samples will contribute to the analysis as the bacterial shedding.
  In EOT/ET visit, blood samples for bacterial shedding will be collected.
SGN1 level in urine for bacterial shedding. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 2, urine samples will be collected for Bacterial Shedding.
  For the first SGN1 administration (C1D1), urine sampling will be conducted within 2 hours before intratumoral injection, 3 hours ±1 hour, 6 hours ±1 hour, 24 hours ±3 hours, 48 hours ±3 hours and 72 hours ±3 hours after end of intratumoral injection.
  For the second and third administration(C1D8 and C1D15),urine samples for bacterial shedding will be collected within 2 hours prior to the start of SGN1 intratumoral injection, and within 24 ± 3 hours after the end of each SGN1 intratumoral injection.
  In EOT/ET visit, urine samples for bacterial shedding will be collected.
SGN1 level in saliva for bacterial shedding. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 2, saliva samples will be collected for Bacterial Shedding.
  For the first SGN1 administration (C1D1), saliva sampling will be conducted within 2 hours before intratumoral injection, 3 hours ±1 hour, 6 hours ±1 hour, 24 hours ±3 hours, 48 hours ±3 hours and 72 hours ±3 hours after end of intratumoral injection.
  For the second and third administration(C1D8 and C1D15),saliva samples for bacterial shedding will be collected within 2 hours prior to the start of SGN1 intratumoral injection, and within 24 ± 3 hours after the end of each SGN1 intratumoral injection.
  In EOT/ET visit, saliva samples for bacterial shedding will be collected.
SGN1 level in feces for bacterial shedding. | Before the first administration up to 28 days after the last dosing.
  In Part 1 and Part 2, feces samples will be collected for Bacterial Shedding.
  For the first SGN1 administration (C1D1), feces sampling for bacterial shedding will be collected by the patient before the intratumoral injection of SGN1,this sample may be collected at any time during the screening period. Additional feces samples will be collected after the end of the intratumoral injection on C1D1 within the time frames below:
  0-24 hours 24-48 hours 48-72 hours
  For the second and third administration(C1D8 and C1D15),feces samples for bacterial shedding will be collected by the patient within 24 hours prior to the start of each SGN1 intratumoral injection, and within 24 hours after the end of each SGN1 intratumoral injection.
  In EOT/ET visit, feces samples will be collected by the subject within 24 hours prior to the EOT/ET visit.
Proinflammatory cytokines | Within 7 days prior to first dosing, and at 2, 4, 6, and 24 hours post end of first infusion.
  Blood samples will be collected to assess proinflammatory cytokines including IL-1β, IFN-γ, TNF-α, IL-6 and IL-8.
Assessment of tumor colonization | From signing the informed consent form until 28 days after the last dose.
  For superficial tumors, biopsy puncture tissue samples or tissue samples within the last half year will be collected from patients (if lesions are appropriate and patients agree) during the screening period, and tissue samples will be collected, and after the intratumoral injection, tissue biopsy puncture will be performed in pre-dose of the C2D15 (within 2 days).

OTHER OUTCOMES:
Expression changes of tumor immune microenvironment related indicators in tumor tissue | From signing the informed consent form until 28 days after the last dose.
  The changes before and after treatment of tumor immune microenvironment related indicators.

CONTACTS AND LOCATIONS:
Locations (4):
- China (2):
  - Guangdong Clifford Hospital, Guangzhou, Guangdong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
- Taiwan (2):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No